CLINICAL TRIAL: NCT03826979
Title: PILATES METHOD ON THE UPPER LIMBS FUNCTIONALITY OF THE MASTECTOMIZED WOMEN
Brief Title: PILATES METHOD ON THE UPPER LIMBS FUNCTIONALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Raphael do Nascimento Pereira, Raphael do Nascimento Pereira, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.510.081
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Breast Neoplasm Female
Keywords: Breast cancer.; Exercise Therapy; Modified Radical Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The participants undergo to a physical therapy rehabilitation program through the Pilates Method for 2 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilates treatment (Experimental): The participants undergo to a physical therapy rehabilitation program through the Pilates Method for 2 months.
  Interventions: Other: Pliates method treatment

INTERVENTIONS:
Other: Pliates method treatment — The participants undergo to a physical therapy rehabilitation program through the Pilates Method for 2 months.

SUMMARY:
INTRODUCTION: Breast cancer is one of the pathologies affecting women worldwide, with a high mortality rate of 14,206 per 100,000 women per year. However, Pilates was used as a therapeutic treatment for women who underwent a modified radical mastectomy, being associated with the alterations when in the postoperative sequels.

OBJECTIVE: to evaluate the Pilates Method in the functionality of women submitted to modified radical mastectomy.

METHOD: This is a quantitative clinical trial, in the form of women included in the project, to undergo a physical therapy rehabilitation program through the Pilates Method for 2 months, where they were evaluated before and after the procedure for measurement and comparison obtained.

CONCLUSION: In this way, the pilates method is presented as an instrument used for the rehabilitation of mastectomized women.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, between 30 and 65 years, with a diagnosis of breast cancer, who underwent radical-mastectomy surgery and who had after 30 postoperative days

Exclusion Criteria:

* Women who present alterations in healing, severe pain, who have another type of treatment, people who lack more than three times in the research, quitters, people with relapses and who do not tolerate the treatment protocol.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women in post-operative radical-mastectomy treatment.
Enrollment: 22 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 months
  Medical Research Council scale for muscle power
Range of motion | 2 months
  Range of motion evaluation by goniometry
Functionality assess with Functional independence measure scale | 2 months
  Functional independence measure scale

CONTACTS AND LOCATIONS:
Locations (1):
- Raphael Pereira, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided